CLINICAL TRIAL: NCT01518738
Title: Attention Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SE-2011-0123
Record Dates: First submitted 2012-01-13; First posted 2012-01-26 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Attention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- breath attention training (Experimental)
  Interventions: Behavioral: breath attention training
- working memory attention training (Active Comparator)
  Interventions: Behavioral: working memory attention training
- no training (No Intervention)

INTERVENTIONS:
Behavioral: breath attention training — 4 week training
  Arms: breath attention training
Behavioral: working memory attention training — 4 week training
  Arms: working memory attention training

SUMMARY:
The purpose of this study is to understand whether attention training is effective in moderating mind wandering.

DETAILED DESCRIPTION:
Our subjective worlds are built from those things in our internal and external environments that capture our attention. Environments can be ambiguous with respect to which objects are most important for our attention, and the characteristics of stimuli that allow them to dominate attention are thus of great interest. Self-relevant objects, such as internally generated experience (e.g. thought), may receive substantial attention, but research on this dimension has been hampered by the difficulty of measuring such objects experimentally. The proposed study seeks to make headway in this area using several behavioral (accuracy, response time, response pattern) measures, with the hypothesis that internally generated experience will vie for attention in a way reflected by behavior. Such research will extend previous work the investigators' lab has done studying stimulus parameters that influence attention, and as a whole may present a more complete picture of how objects and attention interact to shape our worlds.

ELIGIBILITY:
Exclusion Criteria:

* Non-English speakers

Inclusion Criteria:

* Must be able to use a computer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
change in mind wandering frequency after intervention | before intervention and up to 100 weeks later
  mind wandering will be assessed with self-report to intermittent queries such as "just now, was your attention on the present task or unrelated concerns?" Frequency of endorsement will serve as a measure of frequency of mind wandering (ranging in units from 0 - 100% of the time).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Davidson, PhD, Principal Investigator — University Wisconsin Madison
Locations (1):
- University of Wisconsin Brogden Psychology Building, Madison, Wisconsin, United States